CLINICAL TRIAL: NCT06838520
Title: A Prospective Study on the Impact of Androgen Deprivation Therapy (ADT) and Androgen Receptor Pathway Inhibitors (ARPI) on Bone Loss in Prostate Cancer Patients
Brief Title: Effect of ADT and ARPI on Bone Loss of Patients with Prostate Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Bianjiang Liu, Professor, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 2024-SR-999
Record Dates: First submitted 2025-02-03; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: prostate cancer; ADT; ARPI; bone health
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: ADT alone: Men with locally advanced prostate cancer or metastatic hormone-sensitive prostate cancer, about to start treatment.
  ADT including LHRH agonist and antagonist.
  Interventions: Other: Bone health assessment
- Group B: ADT + ARPIs: Men with locally advanced prostate cancer or metastatic hormone-sensitive prostate cancer, about to start treatment.
  ADT including LHRH agonist and antagonist. ARPIs including Abiraterone Acetate, Enzalutamide, Apalutamide, Darolutamide or Rezvilutamide.
  Interventions: Other: Bone health assessment

INTERVENTIONS:
Other: Bone health assessment — Assessments of physical function, DXA scan

SUMMARY:
This study aims to assess the impact of Androgen Deprivation Therapy (ADT) and Androgen Receptor Pathway Inhibitors (ARPI) on bone quality in patients with prostate cancer. Patients undergoing ADT for prostate cancer often experience adverse effects such as decreased bone density and increased fracture risk. While ARPIs are emerging as novel therapeutic agents, their effects on bone quality remain unclear. This study will compare patients receiving combined ADT and ARPI therapy with those receiving ADT alone, evaluating changes in bone density, bone microarchitecture, and bone metabolic markers. The findings will help optimize treatment strategies for prostate cancer patients, reduce the risk of osteoporosis, and improve overall quality of life.

DETAILED DESCRIPTION:
Prostate cancer is the second most common malignancy in men worldwide and ranks fifth in cancer mortality among men. In developed countries in Europe and America, it has the highest incidence rate. In recent years, with the development of the social economy, increased life expectancy, changes in lifestyle, and improvements in the level of medical and health care, the incidence of prostate cancer in China is gradually rising, posing a serious threat to the life safety of men. In China, more than half of the patients with newly diagnosed prostate cancer have advanced metastatic disease. The skeleton is the most common site of metastasis in these patients. Metastatic lesions may cause pathological fractures and spinal cord compression. Patients with extensive bone metastasis are prone to fatigue, weight loss, anemia, and in severe cases, even systemic organ failure. Hormonal therapy based on ADT remains the main treatment for advanced prostate cancer, with the goal of reducing or eliminating the promoting effect of androgens on cancer cell growth.

While ADT treatment benefits patients with metastatic prostate cancer, it also leads to numerous side effects, such as cardiovascular diseases, changes in body composition, decreased bone mineral density (BMD), hot flashes, gynecomastia, cognitive decline, fatigue, anemia, and sexual dysfunction. ADT treatment can affect the number and function of osteoblasts and osteoclasts through various pathways, disrupting the balance of bone remodeling and leading to cancer treatment-induced bone loss. Under normal conditions, testosterone can be converted to estradiol via aromatase and bind to the estrogen receptors on the surface of osteoclasts, indirectly regulating these cells. With increasing age, the bioactivity of both testosterone and estrogen declines in normal men, resulting in low-turnover bone metabolic changes and a bone loss rate of 0.5% to 1% per year. In patients undergoing ADT, the levels of testosterone and estrogen decrease more significantly, and the number of osteoclasts increases markedly. Moreover, ADT treatment can reduce muscle mass and increase fat, leading to sarcopenic obesity, which is accompanied by chronic low-grade inflammation throughout the body and disrupts bone homeostasis. ADT may also lower the levels of circulating vitamin D, which not only affects bone mineralization but also has adverse effects on skeletal muscle and prostate cancer itself. Studies have shown that after 12 months of ADT treatment, the median lumbar spine BMD in patients decreased by an average of 3.6%, higher than that in untreated elderly men (0.5% to 1%). The BLADE study (NCT03202381) confirmed that long-term ADT treatment with either Gonadotropin-releasing hormone (GnRH) receptor agonists or antagonists significantly reduces bone quality. In fact, bone loss caused by ADT treatment can also lead to skeletal-related events (SREs), represented by pathological fractures, bone radiotherapy, bone surgery, and spinal cord compression.

ARPIs play a crucial role in the treatment of prostate cancer. Prostate cancer cells often rely on androgens for growth, and ARPIs work by blocking the androgen receptor pathway, thereby inhibiting the proliferation of cancer cells. These inhibitors, such as abiraterone, enzalutamide, and apalutamide, have significantly improved outcomes for patients with advanced prostate cancer, including those with metastatic castration-resistant prostate cancer (mCRPC). By reducing the levels of androgens or blocking their effects, ARPIs may also negatively impact bone quality in patients with prostate cancer. These agents, by reducing androgen levels, may lead to decreased BMD and increased fracture risk.

The impact of combining ADT with ARPIs on bone quality remains unclear. While clinical trial data on ARPIs in nonmetastatic castration-resistant prostate cancer (nmCRPC) have shown mixed results regarding bone health. Further research is needed to fully understand the combined effects of ADT and ARPIs on bone quality. It is essential to gain a deeper understanding of the patterns of osteoporosis to provide most effective bone-protective therapies to prevent the occurrence of SREs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male gender;
2. Histologically or cytologically confirmed prostate cancer;
3. Clinical stage of metastatic hormone-sensitive prostate cancer (mHSPC);
4. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2;
5. Life expectancy ≥ 12 months;
6. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Suffering from double primary malignancies.
2. Having previously received androgen deprivation therapy (ADT) or other pharmacological treatments (e.g., denosumab, bisphosphonates, or corticosteroids).
3. Having osteoporosis at baseline (T-score ≤ -2.5).
4. Having known bone diseases.
5. Having spinal metastases confirmed by imaging (e.g., ECT, MRI, CT, or PSMA PET-CT).
6. Having poor general condition (i.e., ECOG ≥ 4).
7. Having a life expectancy of less than 12 months.
8. Having elevated serum PSA levels (≥4 ng/dL) or testosterone levels (≥50 ng/dL) after 6 months of ADT.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include male patients with locally advanced or metastatic hormone-sensitive prostate cancer (mHSPC) in mainland China. All patients must have visited the urology or oncology outpatient departments of a tertiary hospital and have a pathological confirmation of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
BMD loss measured at lumbar spine | every 6 months, up to 2 years
  Measured by bone densitometry
BMD loss measured at hip | every 6 months, up to 2 years
  Measured by bone densitometry

SECONDARY OUTCOMES:
trabecular bone score (TBS) changes | every 6 months, up to 2 years
  Measured by bone densitometry
major osteoporotic fracture risk | 24 months
  Estimated by Fracture Risk Assessment Tool (FRAX®)

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Third Affiliated Hospital of Soochow University, Changzhou, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bouillon R, Marcocci C, Carmeliet G, Bikle D, White JH, Dawson-Hughes B, Lips P, Munns CF, Lazaretti-Castro M, Giustina A, Bilezikian J. Skeletal and Extraskeletal Actions of Vitamin D: Current Evidence and Outstanding Questions. Endocr Rev. 2019 Aug 1;40(4):1109-1151. doi: 10.1210/er.2018-00126. PMID 30321335
- [Background] D'Andrea S, Martorella A, Coccia F, Castellini C, Minaldi E, Totaro M, Parisi A, Francavilla F, Francavilla S, Barbonetti A. Relationship of Vitamin D status with testosterone levels: a systematic review and meta-analysis. Endocrine. 2021 Apr;72(1):49-61. doi: 10.1007/s12020-020-02482-3. Epub 2020 Sep 3. PMID 32880851
- [Background] Feng W, Guo J, Li M. RANKL-independent modulation of osteoclastogenesis. J Oral Biosci. 2019 Mar;61(1):16-21. doi: 10.1016/j.job.2019.01.001. Epub 2019 Jan 11. PMID 30929797
- [Background] Kokorovic A, So AI, Serag H, French C, Hamilton RJ, Izard JP, Nayak JG, Pouliot F, Saad F, Shayegan B, Aprikian A, Rendon RA. Canadian Urological Association guideline on androgen deprivation therapy: Adverse events and management strategies. Can Urol Assoc J. 2021 Jun;15(6):E307-E322. doi: 10.5489/cuaj.7355. No abstract available. PMID 34127184
- [Background] Bhowmik D, Song X, Intorcia M, Gray S, Shi N. Examination of burden of skeletal-related events in patients naive to denosumab and intravenous bisphosphonate therapy in bone metastases from solid tumors population. Curr Med Res Opin. 2019 Mar;35(3):513-523. doi: 10.1080/03007995.2018.1532884. Epub 2018 Nov 20. PMID 30286662